CLINICAL TRIAL: NCT00472095
Title: Utility of a Diabetes Themed Fotonovela to Encourage Glycemic Control: a Culturally Appropriate Tool for Education in Latinos
Brief Title: Fotonovela for Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UMC 2007-34
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; fotonovela; Latino
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- diabetes fotonovela (Experimental): spanish language comic book describing diabetes care and consequences
  Interventions: Other: Fotonovela
- placebo fotonovela (Placebo Comparator)
  Interventions: Other: Placebo Fotonovela

INTERVENTIONS:
Other: Fotonovela
  Arms: diabetes fotonovela
Other: Placebo Fotonovela
  Arms: placebo fotonovela

SUMMARY:
Diabetes with poor sugar control can lead to blindness, heart attacks, and amputations. Latinos are more at risk for diabetes. A fotonovela is a type of comic book commonly read by Latinos that might be a way to teach them about the risk of high sugars. The researchers will give patients either a fotonovela about diabetes or one with nothing to do with diabetes. Then they will compare how well sugars were controlled afterward in each group. This way they can see if these fotonovelas were useful.

DETAILED DESCRIPTION:
Elevated glucose in diabetics is a risk for amputation, renal failure, coronary artery disease, neuropathy, and blindness. Controlling glucose better as measured by hemoglobin A1c (A1c) reduces risk for these complications. Information itself is often not enough to change behaviors that increase risk for these complications. Latinos in America are particularly at risk for diabetes (DM) and its complications. A fotonovela is a booklet telling a story using photos with superimposed speech bubbles much like an American style comic book. These are commonly read by Latinos. A fotonovela that tells a story about diabetes complications in a culturally appropriate context that emphasized impact on family might help motivate Hispanic patients to control their sugar better. We propose a single-blinded, randomized, controlled trial of a DM themed fotonovela against a non-DM themed fotonovela to assess its effect on glycemia as measured by A1c. After a primary care provider has seen a Latino type 2 diabetic patient, the investigator will consent them then give them an envelope with the DM themed fotonovela or another that is indistinguishable in the sealed envelope. The primary outcome is hemoglobin A1c one month or more after randomization. Secondary outcomes will A1c in the 1-5 month and 6-12 month time period looking for durability of effect. A sample size of 260 allows for a 30% fallout and gives an 80% power to detect a 0.5% change in A1c with a 1.2% standard deviation on that change with a two-tailed alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* A1c> 7.0

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06; Primary Completion 2016-01-29 (Actual); Study Completion 2016-01-29 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 1 year
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: Roger B Mortimimer, MD, Principal Investigator — UCSF-Fresno Medical Education Program, Department of Family Medicine
Locations (3):
- United States (3):
  - Adventist Health Selma, Fresno, California
  - Clinica Sierra Vista, Fresno, California
  - Deran Colegian Ambulatory Care Center, Fresno, California